CLINICAL TRIAL: NCT04354168
Title: Women's mHealth Program: Nthabi Application in Lesotho
Brief Title: Nthabi in Lesotho - Implementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-40268; R21TW011361-01 (NIH)
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Preconception Care
Keywords: mHealth; Lesotho

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nthabi mHealth Application (Experimental): About 20 women from each of the ten district hospitals will be recruited. Each district hospital will have a separate administrative page on the Nthabi server where women will be enrolled with a unique username and password. Upon enrollment, the women will be asked to engage with Nthabi for two months to discuss the relevant content areas they are interested in learning more about.
  Interventions: Behavioral: mHealth Application

INTERVENTIONS:
Behavioral: mHealth Application — Nthabi mHealth Application delivers educational content and recommendations to minimize or eliminate health risks. The content is delivered via the Nthabi application downloaded on an Android phone smartphone. End-users can select from a list of topics relevant to the Lesotho population to engage with the conversational agent, Nthabi, and discuss conditions such as tuberculosis, HIV testing, healthy diet, and family planning.

SUMMARY:
This project will determine how well the mobile health (mHealth) Nthabi application is introduced and used at district hospitals in Lesotho. This will help with measuring the effectiveness of an evidence-based mHealth application in a low-income country. Three factors will be studied when assessing the mHealth application's overall impact: 1) end-user content knowledge 2) pre and post stage of change and 3) system usage. This data will be collected by the mHealth application. End-users will use the mHealth application over a period of two months. Results will be shared with the clinical, health services research, information technology, and policy communities.

DETAILED DESCRIPTION:
Lesotho has second-highest HIV and fifth-highest tuberculosis prevalence rates worldwide, and a maternal mortality rate (1024/100,000) that is among the highest in Africa. As there are only 6.2 nurses and 0.5 physicians per 10,000 people, both about one-third of the African average, there is an enormous need for eHealth systems to assist the clinical care system.

Preconception care is an effort to focus on engaging young women in their health before they become pregnant since many women enter pregnancy at risk for poor outcomes because of preexisting medical conditions or not following evidence-based preventive action. In 2013, the WHO prioritized research that focuses on developing, delivering, and scaling preconception women's health interventions in low and middle-income countries to optimize health and birth outcomes. The WHO emphasized implementation research as the key step in helping to maximize the coverage and uptake of preconception care to enhance the long-term health outcomes for women and their children.

The existing "Gabby" system is a patient-facing, user-friendly, evidence-based, scalable, culturally adaptive, health communication system designed to improve women's health. The investigator's team has developed and tested several Embodied Conversational Agents (ECAs), which are virtual characters designed using expertise from health communication, psychotherapy, social psychology, sociolinguistics, linguistics, and communication theory.

For this project, the investigators will first adapt the existing "Gabby" system to a culturally appropriate mHealth application, called "Nthabi", and second, study the impact of the Nthabi application into district hospitals in Lesotho in partnership with the Lesotho Boston Health Alliance (LeBoHA) using the existing educational infrastructure. The research team will assess the effectiveness of Nthabi based on the periodic stage of change assessments over the two-month implementation, end-user content knowledge, and system usage.

ELIGIBILITY:
Inclusion Criteria:

* Female Resident of Lesotho
* English Speaking
* Have access to an Android smartphone
* Not currently pregnant at time of enrollment

Exclusion Criteria:

-None

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jack, MD, Principal Investigator — Boston University
Locations (1):
- Lesotho Boston Health Alliance, Maseru, Lesotho

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nkabane-Nkholongo E, Mpata Mokgatle M, Bickmore T, Julce C, Thompson D, Jack BW. Change in sexual and reproductive health knowledge among young women using the conversational agent "Nthabi" in Lesotho: a clinical trial. BMC Glob Public Health. 2024 Sep 5;2(1):60. doi: 10.1186/s44263-024-00091-0. PMID 39681895
- [Derived] Nkabane-Nkholongo E, Mpata-Mokgatle M, Jack BW, Julce C, Bickmore T. Usability and Acceptability of a Conversational Agent Health Education App (Nthabi) for Young Women in Lesotho: Quantitative Study. JMIR Hum Factors. 2024 Mar 12;11:e52048. doi: 10.2196/52048. PMID 38470460
- [Derived] Nkabane-Nkholongo E, Mokgatle M, Bickmore T, Julce C, Thompson D, JAck B. Change in Sexual and Reproductive Health Knowledge among Young Women Using the Conversational Agent "Nthabi" in Lesotho: A Clinical Trial. Res Sq [Preprint]. 2023 Dec 28:rs.3.rs-3788533. doi: 10.21203/rs.3.rs-3788533/v1. PMID 38234736

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nthabi mHealth Application
Started | 160
Completed | 138
Not Completed | 22
Not completed — Lost to Follow-up | 22

BASELINE CHARACTERISTICS:
Arm/Group | Nthabi mHealth Application
Number analyzed (Participants) | 138
Age, Customized [Count of Participants; unit: Participants]
  18-20 | 34
  21-23 | 53
  24-26 | 37
  27-28 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Lesotho | 138

OUTCOME MEASURES:

1. Primary Outcome: Change in Preconception Health Knowledge
Description: Change in preconception health knowledge will be assessed by a change in the percentage correct scores between the Pre and Post tests which were developed by the investigator. Higher positive change scores suggest more knowledge about preconception health.
Time Frame: Baseline, 4 weeks
Measure: Number; unit: percentage change pre to post test
Arm/Group | Nthabi mHealth Application
Number analyzed (Participants) | 138
percentage change pre to post test
  Folic acid knowledge | 58.1
  Family planning knowledge | 14.8
  Healthy eating knowledge | 4.3

2. Secondary Outcome: Ease of Use of Nthabi App
Description: This outcome was assessed by responses to a specific question in an investigator developed survey containing 22 questions eliciting responses on a 4-point Likert scale (strongly agree, agree, disagree, and strongly disagree). The higher the percentage of strongly agree or agree responses the more favorable the results.
Time Frame: 4 weeks
Measure: Number; unit: percentage strongly agree or agree
Arm/Group | Nthabi mHealth Application
Number analyzed (Participants) | 138
percentage strongly agree or agree | 98.6

3. Secondary Outcome: Nthabi App Health Education Content Organized and Timely
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Number; unit: percentage strongly agree or agree
Arm/Group | Nthabi mHealth Application
Number analyzed (Participants) | 138
percentage strongly agree or agree | 95.7

4. Secondary Outcome: Able to Complete Tasks Quickly Using Nthabi
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Number; unit: percentage strongly agree or agree
Arm/Group | Nthabi mHealth Application
Number analyzed (Participants) | 138
percentage strongly agree or agree | 95.7

5. Secondary Outcome: Enjoyed Using the Nthabi App
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Number; unit: percentage strongly agree or agree
Arm/Group | Nthabi mHealth Application
Number analyzed (Participants) | 138
percentage strongly agree or agree | 96.4

6. Secondary Outcome: Intend to Keep Using the Nthabi App
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Number; unit: percentage strongly agree or agree
Arm/Group | Nthabi mHealth Application
Number analyzed (Participants) | 138
percentage strongly agree or agree | 92.1

7. Secondary Outcome: The Nthabi App Was Culturally Appropriate
Description: as for outcome 2
Time Frame: 4 weeks
Measure: Number; unit: percentage strongly agree or agree
Arm/Group | Nthabi mHealth Application
Number analyzed (Participants) | 138
percentage strongly agree or agree | 96.4

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Nthabi mHealth Application
All-Cause Mortality (participants affected / at risk) | 0/138
Serious Adverse Events (participants affected / at risk) | 0/138
Other Adverse Events (participants affected / at risk) | 0/138

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT04354168/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/68/NCT04354168/ICF_001.pdf